CLINICAL TRIAL: NCT07089017
Title: Evaluation of the Feasibility of the Medstrom Medical Device in Laparoscopic Radical Colectomy for Colorectal Cancer
Brief Title: Anesthetic Management Guided by the Medstrom Instrument
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Peiqi Wang, professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PLAGH-L03
Record Dates: First submitted 2025-07-12; First posted 2025-07-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Group C (No Intervention): Standard care using separate BIS (target 40-60) + TOF + standard hemodynamic monitoring.
- Experimental:Group T (Experimental): Continuous monitoring using palmar/plantar sensors with real-time display of integrated pain, sedation, and NMB indices guiding anesthesia management.
  Interventions: Device: medstrom仪器

INTERVENTIONS:
Device: medstrom仪器 — In addition to conventional monitoring methods, such as electrocardiography (ECG), bispectral index (BIS), and train-of-four (TOF) monitoring, Medstrom instruments were utilized to assess and monitor the patient's pain, sedation, and muscle relaxation status.
  Arms: Experimental:Group T

SUMMARY:
This clinical trial seeks to evaluate the feasibility of the Medstrom device for integrated real-time monitoring of pain, sedation, and neuromuscular blockade during laparoscopic radical colectomy. By addressing limitations of conventional multi-device monitoring systems-including data conflicts, interpretation delays, and elevated costs-the study examines whether Medstrom can comprehensively assess intraoperative patient status and effectively guide anesthesia management using validated reference metrics.

Key questions being investigated include:

1. Whether Medstrom can concurrently generate reliable pain, sedation, and neuromuscular indices through a single platform, and if these outputs demonstrate significant correlation with gold-standard measures (HRV for pain, BIS for sedation, TOF for neuromuscular blockade);
2. Whether integrated monitoring reduces intraoperative decision latency (e.g., accelerated pain detection) and mitigates inter-device interference (e.g., BIS distortion by neuromuscular agents);
3. Whether Medstrom introduces device-related adverse events (e.g., cutaneous irritation, signal misinterpretation) while potentially reducing anesthesia complications (e.g., respiratory depression, intraoperative awareness).

Researchers will randomize patients undergoing elective laparoscopic radical colectomy into two groups:

1. Group T（Medstrom -guided）:an intervention group receiving continuous multimodal monitoring via Medstrom,
2. Group C (Conventional):a control group undergoing conventional monitoring (BIS + TOF + hemodynamic parameters).

Synchronized data will be captured at eight predefined intraoperative timepoints for correlation analysis between Medstrom-derived indices and conventional metrics.

DETAILED DESCRIPTION:
This prospective randomized controlled trial (RCT) aims to evaluate the feasibility and safety of the integrated Medstrom monitoring system for real-time, comprehensive assessment of pain, sedation level, and neuromuscular blockade (NMB) during laparoscopic radical colectomy. It addresses significant limitations of conventional fragmented monitoring systems, such as data conflicts between independent devices (e.g., BIS for sedation, TOF for NMB, HRV for pain), delayed clinical interpretation, and suboptimal resource utilization.

The Medstrom technology utilizes palmar/plantar PAM sensors to objectively quantify pain via skin conductance peaks (SCP). SCPs are generated by emotional sweating triggered via spinal nociceptive reflexes, offering key advantages: objective pain quantification (SCP amplitude correlates with stimulus intensity), rapid response (within 1-2 seconds to noxious stimuli), resilience against hemodynamic instability, temperature variations, or medications, and the unique capability to simultaneously output validated sedation and neuromuscular indices. This single-device integration aims to replace the need for separate BIS, TOF, and HRV monitors.

The study design involves 45 patients (adjusted for 10% dropout from n=40) aged 18-65 years with ASA physical status I-III and confirmed colon cancer, undergoing elective laparoscopic radical colectomy. Key exclusions include BMI ≥30, significant organ dysfunction, neurological/neuromuscular disorders, and pregnancy. Participants are randomized into two groups:

1. Medstrom-Guided Group (Intervention): Continuous monitoring using palmar/plantar sensors with real-time display of integrated pain, sedation, and NMB indices guiding anesthesia management.
2. Conventional Monitoring Group (Control): Standard care using separate BIS (target 40-60) + TOF + standard hemodynamic monitoring.

A standardized anesthesia protocol is employed for both groups: Induction with Propofol (1.5-2.5 mg/kg) + Sufentanil (0.2-0.4 μg/kg) + Rocuronium (0.6-1.0 mg/kg), and Maintenance with Propofol (4-12 mg/kg/h) + Remifentanil (0.1-0.2 μg/kg/min) + bolus Rocuronium/Sufentanil as needed. Data collection occurs at 8 critical intraoperative timepoints, including intubation, skin incision, pneumoperitoneum, surgical end, and pre/post supplemental sufentanil administration.

The primary endpoints focus on establishing the feasibility and correlation of the Medstrom indices against current gold standards:

• Correlation of Medstrom-Pain vs. HRV (Pearson/Spearman).

Feasibility is defined by statistically significant correlations (p<0.05, adjusted for multiple comparisons using Bonferroni/Dunn-Šidák).

Secondary outcomes include hemodynamic stability (HR/MAP fluctuations), total anesthetic consumption, device-related adverse events (e.g., skin irritation, signal errors), and analysis of interactions between the integrated indices (using SEM/pathway analysis).

The statistical approach is based on a sample size of 40 (calculated for multivariate repeated measures: α=0.05, β=0.1/power=90%, effect size f²=0.15, variable correlation ρ=0.4), increased to N=45 to account for a 10% dropout rate. Analyses include correlation (95% CIs), consistency (Bland-Altman/ICC for agreement), multivariable comparisons (Hotelling's T² for correlated outcomes), and time effects (Linear mixed models with random intercepts).

This study holds innovative significance as the first RCT to validate a single-device, triple-parameter integrated monitoring system (pain, sedation, NMB) specifically in major abdominal surgery. It addresses critical clinical gaps: providing objective pain quantification (replacing subjective hemodynamic interpretation), minimizing device interference issues (e.g., BIS distortion by neuromuscular agents), and enhancing resource efficiency. The potential clinical impact includes reducing the risk of intraoperative awareness/pain recall and establishing a framework for more cost-effective and streamlined anesthesia management.

ELIGIBILITY:
Inclusion Criteria:

* 1. Timeframe & Location: Patients treated at the First Medical Center of the Chinese PLA General Hospital between June 2025 and December 2026.

  2. Age: 18 to 65 years old. 3. Diagnosis: Pathologically confirmed colon cancer requiring laparoscopic radical resection.

  4. Physical Status: American Society of Anesthesiologists (ASA) Physical Status Class I-III.

  5. Informed Consent: Patients who voluntarily participate in the study and provide written informed consent.

Exclusion Criteria:

- 1. Body Mass Index (BMI): BMI ≥ 30 kg/m². 2. Organ Dysfunction: Severe concomitant cardiac, pulmonary, hepatic, or renal dysfunction.

3. Neurological Conditions:

* History of autonomic nervous system disorders.
* Current use of medications affecting autonomic nervous system function.
* History of neuromuscular dysfunction. 4. Pregnancy/Lactation: Pregnant or lactating women. 5. Recent Surgery: History of secondary surgery within the preceding month. 6. Psychiatric/Cognitive Conditions:
* History of psychiatric disorders or cognitive impairment.
* History of psychotropic or narcotic drug abuse.
* Significant communication barriers.

Withdrawal Criteria:

1.Requirement for conversion to open surgery or other significant deviation from the planned laparoscopic approach due to intraoperative findings.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between HRV and the Medstrom Instrument Pain Index | From the beginning to the end of the operation
  The correlation between HRV and the pain index of the Medstrom instrument under sedation and muscle relaxation with Bis maintained at 40-60 and TOF maintained below 90%

SECONDARY OUTCOMES:
Heart rate | From the beginning to the end of the operation
  Heart rate (bpm) at each time point.
The total amount of anesthetic drugs | From the beginning to the end of the operation
  Total amount of relevant narcotic drugs
Interaction of related indicators | From the beginning to the end of the operation
  Whether there is an interaction between the relevant indices
Mean arterial pressure | From the beginning to the end of the operation
  Mean arterial pressure (mmHg) at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Pei qi Wang, Principal Investigator — The Firsst Medical Center ,Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No